CLINICAL TRIAL: NCT02026609
Title: Glutamine Challenge as Predictor of Hepatic Encephalopathy After Transjugular Intrahepatic Portosystemic Shunt (TIPS)
Status: Terminated | Type: Observational
Why Stopped: Lack of patient accrual
Sponsor: University of Arkansas (Other)
Collaborators: Université de Montréal (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Other Study IDs: #135318
Record Dates: First submitted 2013-12-26; First posted 2014-01-03 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Refractory Ascites; Hepatic Hydrothorax; Hepatic Encephalopathy; Cirrhosis
Keywords: TIPS; Hepatic encephalopathy; Oral glutamine challenge; Psychometric tests; Portal hypertension; Cirrhosis
MeSH Terms: conditions — Ascites; Hepatic Encephalopathy; Fibrosis; Hypertension, Portal | interventions — Psychometrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, and PBMCs
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- TIPS: Patients 18-75 year old with refractory ascites or hepatic hydrothorax and cirrhosis, eligible for TIPS placement. All patients will have a baseline oral glutamine challenge and psychometric tests.
  Interventions: Other: Oral glutamine challenge; Other: Psychometric Tests

INTERVENTIONS:
Other: Oral glutamine challenge — Blood ammonia determination before, 30-, 60-, and 90-minute, after intake of 10 g of L-glutamine
Other: Psychometric Tests — PHES (portosystemic hepatic encephalopathy score) and ICT (inhibitory control test)

SUMMARY:
Transjugular intrahepatic portosystemic shunt (TIPS) is the first-line therapy for patients with cirrhosis and refractory ascites. However, mental changes known as hepatic encephalopathy (HE) frequently occur after TIPS. There is no effective method to predict HE after TIPS. Oral glutamine challenge (OGC) and psychometric tests have been used to assess the risk for HE, but never in patients undergoing TIPS. Severe muscle loss may also predispose patients to HE. The aim of the present study is to assess if both the OGC and psychometric tests can accurately predict the development of overt HE after TIPS. Patients will be studied before TIPS and followed after TIPS for the development of HE. The role of muscle loss in favoring HE, as well as is possible reversibility after TIPS will also be investigated.

DETAILED DESCRIPTION:
In cirrhosis, up to 10% of patients develop refractory ascites. TIPS (transjugular intrahepatic portosystemic shunt) is the first-line therapy for these patients. However, 30% will go on to develop hepatic encephalopathy (HE) as a consequence of TIPS, and there is no effective method to predict this outcome. Oral glutamine challenge (OGC) is used to functionally assess ammonia metabolism, and the severity of porto-systemic collateralization, and it has been used to predict overt HE. Psychometric tests (i.e. Psychometric Hepatic Encephalopathy Score [PHES] and inhibitory control test) allow the identification of covert forms of HE and can also predict overt HE. Severe sarcopenia may also predispose patients to HE. The aim of the present study is to assess if both the degree of impairment in ammonia metabolism as estimated with the OGC, and cognitive status as determined by psychometric tests, can accurately predict the development of overt HE after TIPS. Patients will be studied before TIPS and followed after TIPS for the development of overt HE. The role of sarcopenia in favoring HE, as well as is possible reversibility after TIPS will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis (any etiology)
* Refractory ascites or hepatic hydrothorax and plan for TIPS placement

Exclusion Criteria:

* Well-documented overt hepatic encephalopathy, either persistent or at the time of screening
* Any contraindication for TIPS placement

  * Except for coagulopathy and thrombocytopenia (decided on an individual basis)
* Uncontrolled depression/anxiety disorder or use of antipsychotic drugs
* Active use of alcohol or illicit drugs
* History of dementia
* TIPS planned for another indication.
* Active alcoholic liver disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients will be recruited from the Gastroenterology / Hepatology Clinics at UAMS and other participating centers. Those fulfilling inclusion/exclusion criteria will be invited to participate.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-05; Primary Completion 2015-01-27 (Actual); Study Completion 2015-01-27 (Actual)

PRIMARY OUTCOMES:
Overt hepatic encephalopathy | up to 18 months
  Classified according to West Haven criteria.

SECONDARY OUTCOMES:
Sarcopenia | Baseline and 6 months post-TIPS
  According to CT scan L3 area of muscle mass
Physical activity | Baseline and 6 months post-TIPS
  Pedometer readings and physical activity questionnaire
Dietary Intake | Baseline and 6 months post-TIPS
  Food frequency questionnaire (FFQ, NutritionQuest, Berkeley, CA)

OTHER OUTCOMES:
Skeletal muscle trophic factors | Baseline and 6 months post-TIPS
  IGF-1 and myostatin levels
Glutaminase gene variations | Baseline
  Genetic variations in the glutaminase gene (located at 2q-32-134) consisting of single nucleotide polymorphisms (SNPs) identifying a microsatellite of GCA repeats in the 5' untranslated region
Psychometric tests | 3 and 6 months post-TIPS
  Repeat PHES and ICT

CONTACTS AND LOCATIONS:
Overall Officials: Andres Duarte-Rojo, MD, MSc, Principal Investigator — University of Arkansas
Locations (3):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States
- University of Montreal, Montreal, Quebec, Canada
- University Hospitals of Geneva, Geneva, Switzerland

REFERENCES:
- [Background] Rossle M, Gerbes AL. TIPS for the treatment of refractory ascites, hepatorenal syndrome and hepatic hydrothorax: a critical update. Gut. 2010 Jul;59(7):988-1000. doi: 10.1136/gut.2009.193227. PMID 20581246
- [Background] Romero-Gomez M, Jover M, Del Campo JA, Royo JL, Hoyas E, Galan JJ, Montoliu C, Baccaro E, Guevara M, Cordoba J, Soriano G, Navarro JM, Martinez-Sierra C, Grande L, Galindo A, Mira E, Manes S, Ruiz A. Variations in the promoter region of the glutaminase gene and the development of hepatic encephalopathy in patients with cirrhosis: a cohort study. Ann Intern Med. 2010 Sep 7;153(5):281-8. doi: 10.7326/0003-4819-153-5-201009070-00002. PMID 20820037
- [Background] Romero-Gomez M, Grande L, Camacho I, Benitez S, Irles JA, Castro M. Altered response to oral glutamine challenge as prognostic factor for overt episodes in patients with minimal hepatic encephalopathy. J Hepatol. 2002 Dec;37(6):781-7. doi: 10.1016/s0168-8278(02)00330-6. PMID 12445419
- [Background] Ditisheim S, Giostra E, Burkhard PR, Goossens N, Mentha G, Hadengue A, Spahr L. A capillary blood ammonia bedside test following glutamine load to improve the diagnosis of hepatic encephalopathy in cirrhosis. BMC Gastroenterol. 2011 Dec 8;11:134. doi: 10.1186/1471-230X-11-134. PMID 22151412
- [Background] Duarte-Rojo A, Estradas J, Hernandez-Ramos R, Ponce-de-Leon S, Cordoba J, Torre A. Validation of the psychometric hepatic encephalopathy score (PHES) for identifying patients with minimal hepatic encephalopathy. Dig Dis Sci. 2011 Oct;56(10):3014-23. doi: 10.1007/s10620-011-1684-0. Epub 2011 Apr 3. PMID 21461913
- [Background] Bajaj JS, Saeian K, Verber MD, Hischke D, Hoffmann RG, Franco J, Varma RR, Rao SM. Inhibitory control test is a simple method to diagnose minimal hepatic encephalopathy and predict development of overt hepatic encephalopathy. Am J Gastroenterol. 2007 Apr;102(4):754-60. doi: 10.1111/j.1572-0241.2007.01048.x. Epub 2007 Jan 11. PMID 17222319
- [Background] Tandon P, Ney M, Irwin I, Ma MM, Gramlich L, Bain VG, Esfandiari N, Baracos V, Montano-Loza AJ, Myers RP. Severe muscle depletion in patients on the liver transplant wait list: its prevalence and independent prognostic value. Liver Transpl. 2012 Oct;18(10):1209-16. doi: 10.1002/lt.23495. PMID 22740290